CLINICAL TRIAL: NCT02480413
Title: Evaluation of an Algorithm for Length Based Weight Estimation in Comparison to Already Known Devices Like the Pediatric Emergency Tape (Pädiatrisches Notfalllineal - PNL)
Brief Title: Evaluation of an Algorithm for Length Based Weight Estimation
Status: Completed | Type: Observational
Sponsor: University Children's Hospital, Zurich (Other)
Responsible Party: Principal Investigator, Alexander Schmidt, Dr. med., University Children's Hospital, Zurich
Other Study IDs: KEK-ZH-Nr. 2015-0191 - Part 1
Record Dates: First submitted 2015-06-21; First posted 2015-06-24 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-04

CONDITIONS: Length Based Weight Estimation
Keywords: Broselow Tape; Weight estimation; Patient safety

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Accuracy of an algorithm and the pediatric emergency tape. — No intervention

SUMMARY:
The purpose of this prospective single center study is to investigate if a developed algorithm is more accurate than the pediatric emergency tape (Alpha 1 Werbedesign e.K., Falkenberg, Germany). For this study 500 patients are required to collect anonymized data (length, weight, age, anaesthesia material used during anaesthesia) for achieving a power of 80% during statistical analysis. The main hypothesis ist that the algorithm has a better accuracy than the pediatric emergency tape (53% are in a +/- 10% interval).

DETAILED DESCRIPTION:
This prospective single center study is performed at the university children's hospital zurich. Patients planned for surgery in general anaesthesia with intubation, aged 0 to 16 years and with a body length suitable for the emergency tapes can be included in this study. Patient and parental information is performed during the pre-anaesthetic visit. After written consent the patient will be included. Patient´s length and weight will be measures earliest one day before data collection. Data collection during anaesthesia has no influence on the daily anaesthesia routine and has no impact on patient safety and anaesthesia. Patient's data is made anonymous for further inspection.

Data is documented in Microsoft Excel and statistical analysis calculated with SPSS. 500 patients are needed for a power of 80%. Primary outcome parameter is length-based weight estimation, secondary outcome parameters are length-based age estimation and the correctness of recommended anaesthesia material (endotracheal tube, laryngeal mask, oropharyngeal mask and face mask). Both tools (algorithm and pediatric emergency tape) will be compared with eachother regarding primary and secondary outcome parameters.

ELIGIBILITY:
Inclusion Criteria:

* body length suitable with the investigated emergency tapes
* all patients aged 0 -16 years
* receiving general anaesthesia with intubation

Exclusion Criteria:

* Already included in this study once
* missing patient or parental consent

Ages: 1 Day to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Pediatric patients planned for elecitve surgery in general anaesthesia
Sampling Method: Probability Sample
Enrollment: 492 (Actual)
Dates: Start 2015-07; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
length based weight estimation by algorithm | during anaesthesia

SECONDARY OUTCOMES:
length based age estimation | during anaesthesia
size of endotracheal tube | during anaesthesia
size of laryngeal mask | during anaesthesia
size of facemask | during anaesthesia
size of oropharyngeal tube | during anaesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Alexander R Schmidt, MD, Principal Investigator — University Children´s Hospital Zurich
Locations (1):
- University Childrens Hospital, Zurich, Canton of Zurich, Switzerland